CLINICAL TRIAL: NCT01883310
Title: The Effects of a Task-oriented Circuit Training Combined With Cerebellar Transcranial Direct Current Stimulation on Locomotor Function, Balance and Mobility in Multiple Sclerosis Subjects
Brief Title: Task-oriented Circuit Training Combined With Cerebellar tDCS in Multiple Sclerosis Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOCT_MS_cerebellar tDCS
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis Subjects
Keywords: Multiple Sclerosis; transcranial direct current stimulation; TOCT; task-oriented circuit training; locomotor function; mobility; balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS + TOCT (Active Comparator): The sham transcranial direct current stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 30 s over the right cerebellar position.
  Interventions: Device: sham tDCS + TOCT
- real tDCS + TOCT (Experimental): the real transcranial direct current stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 15 minutes over the right cerebellar position.
  Interventions: Device: real tDCS +TOCT

INTERVENTIONS:
Device: sham tDCS + TOCT — Anodal transcranial direct current stimulation will be delivered through 2 sponge electrodes (surface area: 25 cm2) soaked in a saline solution. For the cerebellar transcranial direct current stimulation, the anodal electrode will be centered on the right cerebellar cortex, 3 cm lateral to the inion, and the cathodal electrode will be positioned on the right buccinator muscle. Anodal stimulation intensity will be set at 2 mili Ampere and delivered using a rechargeable batteries direct current stimulator.The sham transcranial direct current stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 30 s over the right cerebellar position.
  Arms: sham tDCS + TOCT
Device: real tDCS +TOCT — Anodal transcranial direct current stimulation will be delivered through 2 sponge electrodes (surface area: 25 cm2) soaked in a saline solution. For the cerebellar transcranial direct current stimulation, the anodal electrode will be centered on the right cerebellar cortex, 3 cm lateral to the inion, and the cathodal electrode will be positioned on the right buccinator muscle. Anodal stimulation intensity will be set at 2 mili Ampere and delivered using a rechargeable batteries direct current stimulator.The real transcranial direct current stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 15 minutes over the right cerebellar position.
  Arms: real tDCS + TOCT

SUMMARY:
Aims of the study:

This is a double-blind randomized-controlled trial to test the effects of a task oriented training combined with cerebellar transcranial direct current stimulation on locomotor function, mobility and balance in multiple sclerosis subjects with moderate gait impairments (EDSS 4-5,5).

Subjects and methods: 30 multiple sclerosis patients will be recruited in an outpatient rehabilitation clinic University Hospital Ferrara. Informed consent will be obtained. Participants enrolled will included in 2 different treatment groups: Task Oriented Circuit Training (TOCT) + anodal cerebellar transcranial direct current stimulation (experimental group) and TOCT + sham transcranial direct current stimulation over the cerebellum (control group). The group with anodal transcranial direct current stimulation will receive continuous stimulation with intensity of 2 mA during the first 15 minutes of functional circuit training. In the sham session, anodal transcranial direct current stimulation was applied for 30 s and then shut off. Each subject will receive 10 task-oriented training sessions over 2 weeks (5 sessions/week). 3 subjects with a supervisor physiotherapist will take part at the TOCT. During the stimulation sessions both the subject and the researcher, responsible for carrying out clinical tests, will be unaware of the type of stimulation set.

Treatment efficacy outcome measures will be clinical test for gait speed (Timed 25-Foot Walk), walking endurance (six minute walking test), balance (Dynamic Gait Index) and mobility (Time Up and Go Test); self-assessment questionnaire for motor fatigue (Fatigue Severity Scale FSS) and quality of life (Short Form (36) Health Survey).

Outcome measures will be assessed the week prior to treatment initiation (T0), the week after the end of treatment (T1) and at 3 months follow-up (T3) to evaluate treatments retention, by a clinician blinded to the treatment. At the end of each session, the subject will complete a questionnaire where report side effects due to stimulation (headache, neck pain, burning, redness and/or itching in the site of stimulation).

DETAILED DESCRIPTION:
The inclusion criteria will be:

* males and females, community dwelling, age 18 or older;
* diagnosis of multiple sclerosis in a stable phase, which will be defined as a chronic progressive or relapsing-remitting pattern with no relapse during the last 3 months;
* moderate gait impairments referred to Expanded Disability Status Scale between 4 and 5,5 (this EDSS scores refers to people with restricted ambulation who do not need walking aids).

ELIGIBILITY:
Inclusion Criteria:

* males and females, community dwelling, age 18 or older;
* diagnosis of multiple sclerosis in a stable phase, which will be defined as a chronic progressive or relapsing-remitting pattern with no relapse during the last 3 months;
* moderate gait impairments referred to Expanded Disability Status Scale between 4 and 5,5 (this EDSS scores refers to people with restricted ambulation who do not need walking aids).

Exclusion Criteria:

* neurologic conditions in addition to multiple sclerosis that may affect motor function;
* other medical conditions likely to interfere with the ability to safely complete the study protocol;
* impaired cognitive functioning (Mini Mental Status Examination < 24);
* contraindications to transcranial direct current stimulation: intracranial metal implants that can be stimulated, incorrectly positioned or over-heated by the electric current.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline on locomotor function, mobility and balance in multiple sclerosis subjects with gait speed (Timed 25-Foot Walk) | week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)

SECONDARY OUTCOMES:
mobility (Timed Up and Go) | the week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)
Balance (Dynamic Gait Index) | the week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)
walking endurance (six minute walking test | the week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)
fatigue (fatigue severity scale) | the week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)
Short Form (36) Health Survey (SF-36) | the week prior to treatment initiation (T0), the week after the end oftreatment (T1) and at 3 months follow-up (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Nino Basaglia, MD, Principal Investigator — Ferrara University Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No